CLINICAL TRIAL: NCT03465566
Title: Facial Emotion Decoding in Benign Partial Epilepsy of Childhood With Centrotemporal Spikes
Brief Title: Emotion Recognition in Benign Epilepsy of Childhood With Centro-Temporal Spikes (BECTS)
Acronym: BECTS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Alfredo D'Aniello, Medical Doctor, Neurologist and Psychiatrist of child, Principal investigator, Neuromed IRCCS
Other Study IDs: DGN01
Record Dates: First submitted 2018-02-22; First posted 2018-03-14 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: BECTS; Epilepsy, Rolandic
Keywords: Emotion; Social cognition; Childhood epilepsy
MeSH Terms: conditions — Epilepsy, Rolandic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with BECTS: Children with active BECTS according to state-of-the-art diagnostic criteria of ILAE (International League Against Epilepsy). Eligible subjects will be recruited at their first clinical observation in the epilepsy centers involved in the study.
  All subjects will perform five diagnostic evaluations named:
  IDS (Intelligence and Development Scale) MMSPE (Mini Mental State Pediatric Examination) CDI 2 (Children Depression Inventory 2) CBCL (Child Behavior Check List) Tests of facial expression evaluation
  Interventions: Diagnostic Test: IDS;MMSPE;CDI 2;CBCL;tests of facial expression evaluation
- Healthy children: Healthy controls matched for sex, age range, and education with no family history for epilepsy or other neuropsychiatric disorders.
  All subjects will perform the following tests:
  MMSPE (Mini Mental State Pediatric Examination) CDI 2 (Children Depression Inventory 2) CBCL (Child Behavior Check List) Tests of facial expression evaluation
  Interventions: Diagnostic Test: IDS;MMSPE;CDI 2;CBCL;tests of facial expression evaluation

INTERVENTIONS:
Diagnostic Test: IDS;MMSPE;CDI 2;CBCL;tests of facial expression evaluation — Five pictures (including nonfacial features; i.e., hairs) were used for each emotion, giving a total of 25 trials.Stimuli consist of pictures of facial affect taken from the Ekman and Friesen series.

SUMMARY:
The social processes depend on complex cognitive mechanisms, which involve mainly the frontal and temporal lobe regions. Patients with early onset frontal and temporal lobe lesions might later develop important deficits in social integration. Accordingly, children with early onset temporal lobe epilepsy (TLE) demonstrate altered emotion recognition.

DETAILED DESCRIPTION:
Study design: Multicentre, Case-control study.

Emotion recognition is a first step for the development of the capacity to judge the thoughts, intentions, and desires of others. In infants, the capacity to identify, distinguish, and interpret emotions is limited, but these processes are developing rapidly and innately during the first years of life, on the same neural bases as those described in adulthood. Children with BECTS show altered social behavior. In fact, deficit in social cognition could derive from brain dysfunction in the frontotemporal regions primarily affected in BECTS, since these regions are also viewed as playing an important role in social cognition and development of social skills.

The investigators hypothesized that children with BECTS might have altered social cognitive skills and underlying neural networks.

ELIGIBILITY:
Inclusion Criteria:

* children diagnosed with active BECTS (e.g. having at least one seizure with epileptiform abnormalities at EEG)
* treated or not with anti-epileptic drugs; age range between 6 and 11
* infants who have not presented an epileptic seizure within 48 hours before the psychodiagnostic evaluation
* patients with a sleep EEG recording; MMSPE (Mini Mental State Pediatric Examination) ≥23.3

Exclusion Criteria:

* mental retardation
* presence of other neurological or severe neuropsychiatric disorders
* atypical EEG pattern (awake or asleep)

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Two samples matched for number of partecipants, sex, age range, and education. The two samples will include 200 children with BECTS diagnosis, as many healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Number (total amount) of errors in facial emotion recognition | an average of 1 year
  A neuropsychologist will sign the number of errors in recognizing each facial emotion expression
Rating of the intensity of facial expressions | an average of 1 year
  A neuropsychologist will ask the subjects to rate (on a scale from 0 = not at all to 5 = very much) each stimulus with respect to the prototypical expression of that emotion
Rating of the arousal of facial expressions | an average of 1 year
  A neuropsychologist will ask the subjects to evaluate arousal in terms of feeling of high-low energy/wakefulness/alertness by rating each stimulus on a 9-point scale.
Rating of the valence of facial expressions | an average of 1 year
  A neuropsychologist will ask the subjects to evaluate valence in terms of feeling of high-low pleasantness-unpleasantness by rating each stimulus on a 9-point scale.

SECONDARY OUTCOMES:
EEG abnormality lateralization and facial emotion recognition | an average of 1 year
  The investigators will include in statistical analysis the side (dominant hemisphere vs. non-dominant) of EEGraphic abnormalities on awake/sleep recordings

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Di Gennaro, MD, PhD, Study Director — IRCCS Neuromed
Locations (1):
- IRCCS Neuromed, Pozzilli, Isernia, Italy

REFERENCES:
- [Background] De Risi M, Di Gennaro G, Picardi A, Casciato S, Grammaldo LG, D'Aniello A, Lanni D, Meletti S, Modugno N. Facial emotion decoding in patients with Parkinson's disease. Int J Neurosci. 2018 Jan;128(1):71-78. doi: 10.1080/00207454.2017.1366475. Epub 2017 Aug 28. PMID 28796560
- [Background] Meletti S, Picardi A, De Risi M, Monti G, Esposito V, Grammaldo LG, Di Gennaro G. The affective value of faces in patients achieving long-term seizure freedom after temporal lobectomy. Epilepsy Behav. 2014 Jul;36:97-101. doi: 10.1016/j.yebeh.2014.05.002. Epub 2014 Jun 2. PMID 24892756